CLINICAL TRIAL: NCT05534581
Title: Single Shot Pulmonary Vein Isolation: Comparison of Cryoballoon vs. Pulsed Field Ablation in Patients With Symptomatic Paroxysmal Atrial Fibrillation - A Multi-Center Non-Inferiority Design Clinical Trial (The SINGLE SHOT CHAMPION Trial)
Brief Title: SINGLE SHOT CHAMPION
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-D0024
Record Dates: First submitted 2022-08-22; First posted 2022-09-09 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Pulmonary vein isolation; Cryoballoon; Pulsed field ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arctic Front Cryoballoon (Medtronic) (Active Comparator): Pulmonary vein isolation using the Arctic Front Cryoballoon (Medtronic)
  Interventions: Device: PVI using the Arctic Front Cryoballoon (Medtronic)
- Pulsed Field Ablation (FARAPULSE) (Active Comparator): Pulmonary vein isolation using the FARAPULSE PFA system (Boston Scientific)
  Interventions: Device: PVI using FARAPULSE Pulsed Field Ablation (Boston Scientific)

INTERVENTIONS:
Device: PVI using the Arctic Front Cryoballoon (Medtronic) — Patients randomized to the Arctic Front cryoballoon group will undergo PVI using the Arctic Front Cryoballoon (Medtronic). At the end of the procedure, an implantable cardiac monitor will be implanted for the purpose of continuous arrhythmia monitoring.
  Arms: Arctic Front Cryoballoon (Medtronic)
Device: PVI using FARAPULSE Pulsed Field Ablation (Boston Scientific) — Patients randomized to the Pulsed Field Ablation group will undergo PVI using the FARAPULSE PFA system (Boston Scientific). At the end of the procedure, an implantable cardiac monitor will be implanted for the purpose of continuous arrhythmia monitoring.
  Arms: Pulsed Field Ablation (FARAPULSE)

SUMMARY:
Pulmonary vein isolation (PVI) is an effective treatment for atrial fibrillation (AF). Currently, Medtronic Arctic Front Cryoballoon is the most frequently used single shot technology and hence is the benchmark for upcoming technologies. A novel method, pulse-field ablation (PFA) using the FARAPULSE catheter, has recently been introduced (FARAPULSE PFA, Boston Scientific). However, whether FARAPULSE PFA provides effectiveness similar to the standard-of-practice Medtronic Arctic Front Cryoballoon is yet to be investigated. Given that FARAPULSE PFA has shown in studies not to cause any of the severe complications reported in association with traditional PVI while being highly effective, it might be even safer and more effective for use in AF ablation procedures.

The aim of this trial is to compare the efficacy and safety of PVI using FARAPULSE PFA (Boston Scientific) and the Arctic Front Cryoballoon (Medtronic) in patients with symptomatic paroxysmal AF undergoing their first PVI.

This is an investigator-initiated, multicenter, randomized controlled, open-label trial with blinded endpoint adjudication. Given that the Medtronic Arctic Front Cryoballoon is the standard-of-practice for PVI and the FARAPULSE PFA is the novel technology, this trial has a non-inferiority design.

The null hypothesis with regards to the primary efficacy endpoint is that the FARAPULSE PFA (Boston Scientific) shows lower efficacy compared to the Arctic Front Cryoballoon (Medtronic) and that therefore more episodes of first recurrence of any atrial arrhythmia between days 91 and 365 will be observed in patients with symptomatic paroxysmal AF undergoing their first PVI. Hence, the alternative hypothesis postulates that the FARAPULSE PFA is non-inferior to the Arctic Front Cryoballoon. Rejection of the null hypothesis is needed to conclude non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation documented on a 12 lead ECG or Holter monitor (lasting ≥30 seconds) within the last 24 months. According to current guidelines, paroxysmal is defined as any AF that converts to sinus rhythm within 7 days either spontaneously or by pharmacological or electrical cardioversion
* Candidate for ablation based on current AF guidelines
* Continuous anticoagulation with Vitamin-K-Antagonists or a novel oral anticoagulant for ≥4 weeks prior to the ablation; or a transesophageal echocardiography and/or computer tomography that excludes left atrial (LA) thrombus ≤48 hours before ablation
* Age of 18 years or older on the date of consent
* Informed Consent as documented by signature

Exclusion Criteria:

* Previous left atrial (LA) ablation or LA surgery
* AF due to reversible causes (e.g. hyperthyroidism, cardiothoracic surgery)
* Intracardiac thrombus
* Pre-existing pulmonary vein stenosis or PV stent
* Pre-existing hemidiaphragmatic paralysis
* Contraindication to anticoagulation or radiocontrast materials
* Prior mitral valve surgery
* Severe mitral regurgitation or moderate/severe mitral stenosis
* Myocardial infarction during the 3-month period preceding the consent date
* Ongoing triple therapy
* Cardiac surgery during the three-month interval preceding the consent date or scheduled cardiac surgery/TAVI procedure
* Significant congenital heart defect (including atrial septal defects or PV abnormalities but not including PFO)
* NYHA class III or IV congestive heart failure
* Left ventricular ejection fraction (LVEF) <35%
* Hypertrophic cardiomyopathy (wall thickness >1.5 cm)
* Significant chronic kidney disease (CKD; eGFR <30 ml/min)
* Uncontrolled hyperthyroidism
* Cerebral ischemic event (stroke or TIA) during the six-month interval preceding the consent date
* Ongoing systemic infections
* History of cryoglobulinemia
* Cardiac amyloidosis
* Pregnancy
* Life expectancy less than one (1) year per physician opinion
* Currently participating in any other clinical trial, which may confound the results of this trial.
* Unwilling or unable to comply fully with study procedures and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Time to first recurrence of any atrial tachyarrhythmia | Days 91 to 365 post-ablation
  Time to first recurrence of any atrial tachyarrhythmia (atrial fibrillation [AF], atrial flutter [AFL] or atrial tachycardia [AT]) between days 91 and 365 post ablation as detected on continuous implantable cardiac monitor (ICM). AF, AFL or AT will qualify as a recurrence after ablation if it lasts 120 s or longer on ICM (the minimum programmable episode interval).

SECONDARY OUTCOMES:
Number of participants with complications | Days 0 to 30 post-ablation
  Composite safety endpoint composed of:
  * cardiac tamponade requiring drainage
  * persistent phrenic nerve palsy lasting >24 hours
  * serious vascular complications requiring intervention
  * stroke/TIA
  * atrioesophageal fistula
  * death
Total procedure time | Day 0
  Procedural endpoint
Total left atrium indwelling time | Day 0
  Procedural endpoint
Total fluoroscopy time | day 0
  Procedural endpoint
Total radiation dose | Day 0
  Procedural endpoint
Contrast agent usage | Day 0
  Procedural endpoint
Increase in hsTroponin on day 1 post-ablation | Day 1
  Procedural endpoint
Proportion of isolated veins | Day 0
  Assessed by post-ablation 3D electro-anatomical mapping in the first 25 patients in each study group
Proportion of isolated carinas | Day 0
  Assessed by post-ablation 3D electro-anatomical mapping in the first 25 patients in each study group
Lesion size | Day 0
  Assessed by post-ablation 3D electro-anatomical mapping in the first 25 patients in each study group
Time to first recurrence of atrial tachyarrhythmia between days 1 and 90 after ablation | Days 1 to 90 post-ablation
  Time to first recurrence of any atrial tachyarrhythmia (atrial fibrillation [AF], atrial flutter [AFL] or atrial tachycardia [AT]) between days 1 and 90 post ablation as detected on continuous implantable cardiac monitor (ICM). AF, AFL or AT will qualify as a recurrence after ablation if it lasts 120 s or longer on ICM (the minimum programmable episode interval).
Arrhythmia burden evaluated based on continuous ICM (overall AF burden = % time in AF) | Between: 0-90 days, 91-365 days, 365 days up to 3.5 years
  Assessed by the ICM Core Lab post implantation: between 0-90 days; 91-365 days, 365 days to explantation/end of life of the ICM
Arrhythmia being AF or organized atrial arrhythmias (atrial flutter or atrial tachycardias) | 3, 12, 24 and 36 months follow up
  Comparison of the prevalence of the type of arrhythmia recurrences during follow-up being AF or organized atrial arrhythmias (AFL or AT)
Average heart rates | Months 1, 2 and 3 post-ablation
  Average heart rates in ICM documentation in months 1, 2 and 3 after ablation
Proportion of patients admitted to the hospital or emergency room because of documented recurrence of atrial arrhythmias | Postablation 3 months (+/- 2 weeks), 12 months (+/- 2 months), 24 months (+/- 2 months) and 36 months (+/- 2 months)
  Based on telephone follow-up
Proportion of patients undergoing electrical cardioversion because of documented recurrence of atrial arrhythmias | Postablation 3 months (+/- 2 weeks), 12 months (+/- 2 months), 24 months (+/- 2 months) and 36 months (+/- 2 months)
  Based on telephone follow-up
Proportion of patients undergoing a repeat ablation procedure because of documented recurrence of atrial arrhythmias | Postablation 3 months (+/- 2 weeks), 12 months (+/- 2 months), 24 months (+/- 2 months) and 36 months (+/- 2 months)
  Based on telephone follow-up
Reinitiation of antiarrhythmic drugs during follow-up | Months 3, 12, 24 and 36 post-ablation
  Reinitiation of antiarrhythmic drugs during follow-up based on telephone follow-up
Number of reconnected veins evaluated during redo-procedures | During redo-procedure, expected to be on average 20-60 minutes
Evolution of Quality of Life through months 3 and 12 | Months 3 and 12 post-ablation
  QoL questionnaires (EQ-5D) will be sent to the patients by mail after 3 and 12 months to compare the evolution of QoL after the ablation
Stroke including TIA after 3, 12, 24 and 36 months | Months 3, 12, 24 and 36 post-ablation
Death cardiovascular or non-cardiovascular after 3, 12, 24 and 36 months | Months 3, 12, 24 and 36 post-ablation
Sites (anatomical location) of vein reconnection assessed in study patients undergoing a Redo-Procedure at one of the study centres | During redo-procedure, expected to be on average 20-60 minutes
Size (area calculate in cm2) of antral scar area assessed in study patients undergoing a Redo-Procedure at one of the study centres | During redo-procedure, expected to be on average 20-60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Reichlin, MD, Principal Investigator — Inselspital, Bern University Hospital
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel
  - Inselspital, Bern University Hospital, Bern

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Reddy VY, Neuzil P, Koruth JS, Petru J, Funosako M, Cochet H, Sediva L, Chovanec M, Dukkipati SR, Jais P. Pulsed Field Ablation for Pulmonary Vein Isolation in Atrial Fibrillation. J Am Coll Cardiol. 2019 Jul 23;74(3):315-326. doi: 10.1016/j.jacc.2019.04.021. Epub 2019 May 11. PMID 31085321
- [Derived] Reichlin T, Kueffer T, Badertscher P, Juni P, Knecht S, Thalmann G, Kozhuharov N, Krisai P, Jufer C, Maurhofer J, Heg D, Pereira TV, Mahfoud F, Servatius H, Tanner H, Kuhne M, Roten L, Sticherling C; SINGLE SHOT CHAMPION Investigators. Pulsed Field or Cryoballoon Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2025 Apr 17;392(15):1497-1507. doi: 10.1056/NEJMoa2502280. Epub 2025 Mar 31. PMID 40162734